CLINICAL TRIAL: NCT02684435
Title: Contrast-enhanced Ultrasound for Complex Kidney Lesion Diagnosis in Patients With CKD (CEUS CKD)
Brief Title: Contrast-enhanced Ultrasound of the Kidney
Acronym: CEUS-CKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Vanderbilt University (Other); North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-1866
Record Dates: First submitted 2016-02-03; First posted 2016-02-18 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-04

CONDITIONS: Chronic Kidney Disease; Cystic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases, Cystic | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perflutren lipid microsphere (Experimental): Activate by shaking for 45 seconds using VIALMIX. Use activated product within 5 minutes. Infusion: The recommended infusion dose for activated perflutren is via an IV infusion of 1.3 mL added to 50 mL of preservative-free saline. The rate of infusion should be initiated at 4.0 mL/minute, but titrated as necessary to achieve optimal image enhancement, not to exceed 10 mL/minute per P.I. approval
  Interventions: Drug: Perflutren lipid microsphere

INTERVENTIONS:
Drug: Perflutren lipid microsphere — Dosing per approved package label
  Other Names: Definity®; Microbubble contrast agent

SUMMARY:
The purpose of this research study is to evaluate contrast-enhanced ultrasound for kidney malignancies

DETAILED DESCRIPTION:
This is an investigator-initiated, prospective study designed to evaluate the accuracy of contrast-enhanced ultrasound (CEUS) with microbubble contrast agent (perflutren lipid; Definity®) to identify malignancy in patients with kidney disease, a known risk factor for kidney malignancy, in whom a conventional ultrasound (US) shows an indeterminate cystic kidney lesion.

The primary objective of the study is to estimate the sensitivity of CEUS in diagnosing kidney malignancy in patients with a risk factor for kidney malignancy and compare it to the current gold standard test in this patient population. Secondary analysis will include more optimal contrast-enhanced imaging with computed tomography (CT) or magnetic resonance imaging (MRI) in a subset of patients who can receive these studies. The study outcome will lead to immediate clinical application in patients with chronic kidney disease. Given the cost-effectiveness and adverse event profile, it has excellent potential to become established as first line diagnostics in the general patient population as well.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the present study, patients must meet the following criteria:

1. Able to provide written informed consent
2. Willing to comply with protocol requirements
3. At least 18 years of age
4. Have kidney disease, defined as either CKD II-VI, determined by estimated glomerular filtration rate (GFR) of <90 and derived from serum creatinine measurements, or albuminuria/proteinuria, determined by albumin to creatinine ratio or protein to creatinine ratio of >30mg/gm, or having received a kidney transplant
5. Have at least one kidney lesion identified but incompletely characterized on a non-contrasted US, CT, or MR exam for which the patient's provider recommends follow-up studies or further evaluation with an additional imaging tests.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded for enrollment:

1. Critically ill or medically unstable and whose critical course during the observation period would be unpredictable (e.g., chronic obstructive pulmonary disease (COPD) requiring oxygen)
2. Known hypersensitivity to sulfur hexafluoride or to any component of perflutren lipid (Definity®)
3. Right to left shunt, severe pulmonary hypertension (Pulmonary artery pressure >90mmHg), or adult respiratory distress syndrome
4. Active cardiac disease including any of the following:

   * Severe congestive heart failure (class IV in accordance with the classification of the New York Heart Association)
   * Unstable angina.
   * Severe arrhythmia (i.e. ventricular tachycardia, flutter fibrillation; ventricular premature complexes occurring close to the preceding T- wave, multifocal complexes).
   * Myocardial infarction within 14 days prior to the date of proposed Definity® administration.
   * Uncontrolled systemic hypertension (systolic blood pressure (BP) >180 mm Hg and/or diastolic BP >100 mm Hg despite optimal medical management
5. Is in an intensive care setting
6. Has an unstable neurological disease (e.g cerebrovascular accident (including transient ischemic attacks (TIAs) within the 3 months before signing of informed consent
7. Has undergone an invasive procedure on kidney lesion (e.g. tissue biopsy, surgery, nonsurgical cytoreductive procedure) since identification of lesion via US without contrast
8. Has any other medical condition or other circumstances that would significantly decrease the chances of obtaining reliable data or of achieving the study objectives such as:

   * Mental illness
   * Drug abuse
9. Female patient who is pregnant or lactating (the possibility of pregnancy has to be excluded by negative serum or urine beta human chorionic gonadotropin results, obtained within 24 hours before the perflutren lipid administration, or on the basis of patient history, e.g.: tubal ligation, hysterectomy or a minimum of 1 year without menses)
10. Obesity that limits obtainment of acceptable images

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-02; Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Chang, M.D., Principal Investigator — University of North Carolina Kidney Center 7024 Burnett Womack CB #7155 Chapel Hill, NC 27599-7155
Locations (2):
- United States (2):
  - University of North Carolina of Chapel hill, Chapel Hill, North Carolina
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maisonneuve P, Agodoa L, Gellert R, Stewart JH, Buccianti G, Lowenfels AB, Wolfe RA, Jones E, Disney AP, Briggs D, McCredie M, Boyle P. Cancer in patients on dialysis for end-stage renal disease: an international collaborative study. Lancet. 1999 Jul 10;354(9173):93-9. doi: 10.1016/s0140-6736(99)06154-1. PMID 10408483
- [Background] Lindner JR. Microbubbles in medical imaging: current applications and future directions. Nat Rev Drug Discov. 2004 Jun;3(6):527-32. doi: 10.1038/nrd1417. No abstract available. PMID 15173842
- [Background] Lind Ramskov K, Thomsen HS. Nephrogenic systemic fibrosis and contrast medium-induced nephropathy: a choice between the devil and the deep blue sea for patients with reduced renal function? Acta Radiol. 2009 Nov;50(9):965-7. doi: 10.3109/02841850903209218. No abstract available. PMID 19863403
- [Background] Nicolau C, Bunesch L, Pano B, Salvador R, Ribal MJ, Mallofre C, Sebastia C. Prospective evaluation of CT indeterminate renal masses using US and contrast-enhanced ultrasound. Abdom Imaging. 2015 Mar;40(3):542-51. doi: 10.1007/s00261-014-0237-3. PMID 25209216
- [Background] Ascenti G, Mazziotti S, Zimbaro G, Settineri N, Magno C, Melloni D, Caruso R, Scribano E. Complex cystic renal masses: characterization with contrast-enhanced US. Radiology. 2007 Apr;243(1):158-65. doi: 10.1148/radiol.2431051924. PMID 17392251

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: lesions
Period: Overall Study
Arm/Group | Perflutren Lipid Microsphere
Started | 63; 64 lesions
Completed | 63; 64 lesions
Not Completed | 0; 0 lesions

BASELINE CHARACTERISTICS:
Arm/Group | Perflutren Lipid Microsphere
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 33
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions With a Change in Radiologist's Evaluation
Description: Lesions will be assessed for change in size, calcification, and septation based on Bosniak criteria (I, II, IIF, III, IV) to determine whether a lesion has progressed, regressed, or is stable.
Time Frame: Baseline, 1 year
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Perflutren Lipid Microsphere
Number analyzed (Participants) | 63
Number analyzed (lesions) | 64
lesions | 24

2. Primary Outcome: Sensitivity of Qualitative Interpretations of CEUS in Diagnosing Kidney Malignancy
Description: PRELIMINARY RESULTS of sensitivity of qualitative interpretations of CEUS in diagnosing kidney malignancy in patients with CKD and a suspicious or indeterminate lesion on non-contrasted imaging compared to the truth standard
Time Frame: Baseline, 1 year
Measure: Number; unit: percentage of positive scans
Arm/Group | Perflutren Lipid Microsphere
Number analyzed (Participants) | 63
percentage of positive scans | 75

3. Primary Outcome: Specificity of Qualitative Interpretations of CEUS
Description: PRELIMINARY RESULTS of specificity of qualitative interpretations of CEUS in diagnosing kidney malignancy in patients with CKD and a suspicious or indeterminate lesion on non-contrasted imaging compared to the truth standard
Time Frame: Baseline, 1 year
Measure: Number; unit: percentage of negative scans
Arm/Group | Perflutren Lipid Microsphere
Number analyzed (Participants) | 63
percentage of negative scans | 71

4. Secondary Outcome: Specificity of Quantitative Metrics Generated From CEUS in Diagnosing Kidney Malignancy in Patients With CKD and a Suspicious or Indeterminate Lesion on Non-contrasted Imaging Compared to the Truth Standard
Description: Specificity of Quantitative Metrics Generated From CEUS in Diagnosing Kidney Malignancy in Patients With CKD and a Suspicious or Indeterminate Lesion on Non-contrasted Imaging Compared to the Truth Standard
Time Frame: Baseline, 1 Year
Population: Quantitative analysis unable to be conducted on cystic lesions and required solid portions, so data was not collected
Arm/Group | Perflutren Lipid Microsphere
Number analyzed (Participants) | 0

5. Secondary Outcome: Sensitivity of Quantitative Metrics Generated From CEUS in Diagnosing Kidney Malignancy in Patients With CKD and a Suspicious or Indeterminate Lesion on Non-contrasted Imaging Compared to the Truth Standard
Description: Sensitivity of Quantitative Metrics Generated From CEUS in Diagnosing Kidney Malignancy in Patients With CKD and a Suspicious or Indeterminate Lesion on Non-contrasted Imaging Compared to the Truth Standard
Time Frame: Baseline, 1 Year
Population: Quantitative analysis unable to be conducted on cystic lesions and required solid portions, so data was not collected
Arm/Group | Perflutren Lipid Microsphere
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 30 minutes post imaging at baseline visit
Arm/Group | Perflutren Lipid Microsphere
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 1/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perflutren Lipid Microsphere (N=63)
Bilateral back pain that resolved by the time of discharge. (Musculoskeletal and connective tissue disorders) | 1 (1) — Bilateral back pain that resolved by the time of discharge. Patient also has chronic back issues and some difficulty with mobility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT02684435/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT02684435/ICF_001.pdf